CLINICAL TRIAL: NCT02873052
Title: MyoVista Measurements in Patients With Atherosclerosis and CAD
Status: Completed | Type: Observational
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Heart Test Laboratories, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Other Study IDs: 21562-01
Record Dates: First submitted 2016-06-29; First posted 2016-08-19 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease (CAD); Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cholesterol measurements, Inflammatory markers (Interleukin-6 and C-reactive protein).
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MyoVista — The clinical set up of MyoVista™ is identical to that of a traditional 12-lead ECG but it obtains and processes signal information in a way that permits much greater resolution of the electrical activity associated with the myocardium MyoVista.

SUMMARY:
The MyoVista system is a novel electrocardiogram technology that provides non-invasive assessment of myocardial abnormalities by analyzing energy changes at the cellular level of the myocardium.

DETAILED DESCRIPTION:
The MyoVista iECG Electrocardiograph is a diagnostic device used to process electrical signals transmitted through electrocardiograph electrodes and to detect ischemia abnormalities based on electrical waveform, patient data, demographics, algorithmic sensitivity and software based informatics. The MyoVista provides the clinician with a standard ECG conventional waveform, along with an additional report derived from the proprietary informatics exclusive to the MyoVista.

The device holds a lot of promise for early intervention to properly diagnose and treat patients under risk timely and effectively. The MyoVista captures and amplifies signals from the myocardial tissue. These signals are then processed and compared to an algorithm that looks for certain changes occurring in these processed waveforms. The changes that have been identified occur much sooner than those processed by a traditional electrocardiogram (ECG). These recordings focus on early detection of myocardial abnormalities by non-linear analysis of electrical activity and physiological phenomenon. This novel assessment might be capable of detecting subclinical myocardial dysfunction in a variety of heart diseases.

The study would compare MyoVista results to subclinical measures of atherosclerosis (CAC and CT angiography) in 200 subjects at risk for coronary disease. Correlations between the MyoVista reading and the presence of calcified plaque, soft plaque, CTA stenosis, will be determined.

This study has the potential to confirm MyoVista as a reliable and sensitive marker of atherosclerosis. Findings may provide a strong indication for the value of a MyoVista test to confirm CAD in clinical practice, and for the clinical application of MyoVista in management of coronary disease and atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* From (and inclusive of) ages of 18 to 80 years
* Body mass index (BMI) between 18 and 39.9 (kg/m2)
* Able to lie (supine) still comfortably on the back for at least 20 minutes

Exclusion Criteria:

* Known history of cancer, other than non-melanoma skin cancer
* Known history of heart disease or heart rhythm abnormalities
* Known history of cardiovascular disease
* Known history of Peripheral Artery Disease (PAD)
* Known history of claudication
* History of amputation or loss of limb(s)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac CT for clinical reasons in the outpatient center.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
Ability of MyoVista to measures subclinical atherosclerosis | 5 Months

CONTACTS AND LOCATIONS:
Overall Officials: Tess Jackovich, Study Director — VP-Business Development
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be tabulated and analysed. Study site will not share any of the subject identifiers.